CLINICAL TRIAL: NCT05397743
Title: A Prospective Study About Global, Psychological and Visual Quality of Life After an Eye Surgical Removal (Enucleation or Evisceration)
Brief Title: Quality Of Life After Eye Surgical Removal
Acronym: QOLAE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2022/673
Record Dates: First submitted 2022-05-18; First posted 2022-05-31 (Actual); Last update posted 2022-07-26 (Actual); Status verified 2022-07

CONDITIONS: Evisceration; Traumatic, Eye
Keywords: Enucleation
MeSH Terms: interventions — Quality of Life

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Questionnaires (Experimental): Questionnaires for global, psychological and visual Quality of Life (QoL)
  Interventions: Other: Quality of Life

INTERVENTIONS:
Other: Quality of Life — Questionnaire Perceived stress scale (PSS) + Questionnaire Short form 36 (SF-36) + Questionnaire Visual functioning questionnaire 25 (VFQ-25)

SUMMARY:
Studies have shown that health-related quality of life (HRQOL) was worse among patients who underwent surgical eye removal compared to the general population in Denmark.

A third of eye amputated patients suffered from anxiety and depression. Most of the available evidence on the subject is based on retrospective studies that interviewed patients several years after surgery, which can potentially introduce biases.

Moreover, in the literature, there are no data concerning postoperative psychological and visual impact.

ELIGIBILITY:
Inclusion Criteria:

* Patient who underwent an eye removal surgery: evisceration, enucleation or exenteration

Exclusion Criteria:

* Patient who underwent bilateral eye removal surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-05-23 (Actual); Primary Completion 2023-08-23 (Estimated); Study Completion 2023-08-23 (Estimated)

PRIMARY OUTCOMES:
Score VFQ 25 score up to 3 months after surgery | Month 3
  100 = Best score, 0 = Worst possible score

SECONDARY OUTCOMES:
PSS score up to 3 months after surgery | Month 3
  * score from 0 to 13 = low stress
  * score from 14 to 26 = moderate stress
  * score from 27 to 40 = high perceived stress.
SF-36 score up to 3 months after surgery | Month 3
  The SF-36, as described in the name, is a 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state

CONTACTS AND LOCATIONS:
Overall Officials: Lauriana SOLECKI, MD, Principal Investigator — CHU de Besançon
Locations (1):
- CHU de Besançon, Besançon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasmussen ML, Ekholm O, Prause JU, Toft PB. Quality of life of eye amputated patients. Acta Ophthalmol. 2012 Aug;90(5):435-40. doi: 10.1111/j.1755-3768.2010.02092.x. Epub 2011 Feb 10. PMID 21310012
- [Background] Ahn JM, Lee SY, Yoon JS. Health-related quality of life and emotional status of anophthalmic patients in Korea. Am J Ophthalmol. 2010 Jun;149(6):1005-1011.e1. doi: 10.1016/j.ajo.2009.12.036. Epub 2010 Mar 15. PMID 20231012
- [Background] Damato B. Improving the quality of life of patients undergoing enucleation. Eye (Lond). 2022 Aug;36(8):1711. doi: 10.1038/s41433-021-01783-9. Epub 2021 Oct 13. No abstract available. PMID 34645962